CLINICAL TRIAL: NCT04972409
Title: Value of Information of Secondary dAta in ONCOGEnetics
Acronym: VISAGE-ONCO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Georges Francois Leclerc (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-A02303-54
Record Dates: First submitted 2021-06-28; First posted 2021-07-22 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2021-07

CONDITIONS: Cancer; Genetic Predisposition; Secondary Fundings
MeSH Terms: conditions — Neoplasms; Genetic Predisposition to Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
VISAGE-ONCO study is a qualitative transversal study aiming to identify and describe processes and mechanisms that explain in cancerology the feelings and experience of patients and health professionals with regard to the possibility of having access to secondary findings generated by the use High-speed exome sequencing . Semi-structured interviews will be conducted with patients and health professionals to answer this aims from 2 situations.

The first situation is in the context of the standard practice for theranostic purposes, where somatic and constitutional analysis of the various genes involved in carcinogenesis is carried out systematically in parallel. Patients are informed that the analysis of these genes may reveal the existence of a genetic predisposition to another type of cancer than the one for which patients have consulted, with a risk for themselves or their relatives, which could modify their management. This targeted information on genetic predisposition genes to cancer is therefore provided as part of standard management for theranostic purposes, but without any detailed exploration of the reasons why patients wanted to be informed.

The second situation is in the framework exome analysis position in the strategy of genetic redisposition factors identification in early-onset cancer study (EX²TRICAN NCT04141462) where all the genes identified in human pathology are part of the analysis. Patients have the possibility of accessing a result concerning a gene that may or may not be linked to a hereditary cancer risk if patients have ticked off in the consent form the wish to be informed.

Therefore, two distinct questions arise:

* That of understanding the wish of patients to be given back actionable data which can be identified in a fortuitous way within the framework of standard management for theranostic purposes and in EX²TRICAN, by taking into account the fact that these data can constitute an opportunity for the patient in terms of management; but patients also constitute a risk of transmission for they relatives, and a psychological risk by the anxiety generated;
* The wish to have access - or not - to data which are not actively sought today within the framework of standard care for theranostic purposes and in EX²TRICAN (genetic alterations increasing the risk of cardiovascular or metabolic diseases), but which could be proposed in a systematic way in the future because of their actionable character.

ELIGIBILITY:
Inclusion Criteria:

Standard care patients for theranostic goal

* Histological or cytological evidence of a diagnosis of metastatic or locally advanced solid tumor
* Tumor material available and usable for the analyses required by the study
* Request for genetic analysis to be performed at the initiation of the 1st or 2nd line of treatment
* Normal biological parameters
* Life expectancy ≥ 6 months
* Performance status ≤ 1
* Social security affiliation
* Who have received information and agreed to participate

Patient from EX²TRICAN study

* Histological or cytological evidence of a diagnosis of metastatic or locally advanced solid tumor
* Having cancer before age 40
* Patient affiliated to social security
* Availability of a tumor sample if secondary functional studies are required
* Availability of the 2 parents when the trio approach is required
* Availability of affected relatives
* Who have received information and agreed to participate

Health professional

* To be oncologist or geneticist or genetic counselor and able to be inform, prescribe and transmit the results of secondary data
* Working at university hospital center of dijon or cancerology center Georges Francois Leclerc at Dijon
* Who have received information and agreed to participate

Exclusion Criteria:

Standard care patients for theranostic goal

* History of Human immunodeficiency virus infection
* History of Hepatitis B virus /Hepatitis C virus infection
* To be pregnant or likely to be or breastfeeding disorders psychiatric

Patient from EX²TRICAN study

* Minor index cases
* Disorders psychiatric

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cancer who will undergo exomes analysis
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2019-12-09 (Actual); Primary Completion 2022-06-09 (Estimated); Study Completion 2022-12-09 (Estimated)

PRIMARY OUTCOMES:
Patient's experience through semi-structured interviews | 1 day (during the interview)
  Patients were asked during a semi-structured interview, to understand their feelings and experience ith regard to the possibility of having access to secondary findings

CONTACTS AND LOCATIONS:
Overall Officials: François GHIRINGHELLI, PU-PH, Principal Investigator — Centre Georges Francois Leclerc
Locations (1):
- Centre Georges Francois Leclerc, Dijon, France